CLINICAL TRIAL: NCT02153424
Title: Early Post-marketing Study of Eliquis (Apixaban)
Status: Withdrawn | Type: Observational
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-330
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NVAF patients in Mexico treated with Apixaban: All patients with NVAF at the sentinel site for the CNFV in Mexico who received at least 1 dose of Apixaban to reduce the risk of stroke or systemic embolism during the specified 24-month study period
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis

SUMMARY:
The primary objective of the study is to identify and describe any suspected (AEs) in all patients with NVAF treated with Apixaban, as a request of the National Center of Pharmacovigilance (CNFV) in Mexico.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* All patients with NVAF at the sentinel site for the CNFV in Mexico who received at least 1 dose of Apixaban to reduce the risk of stroke or systemic embolism during the specified 24-month study period

Exclusion Criteria:

* Subjects who received Apixaban as part of a clinical trial
* Subjects who received Apixaban for any indication other than local approval (ie, to reduce the risk of stroke and systemic embolism in patients with NVAF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sentinel site for the CNFV in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Determine the reporting rate of on-treatment adverse events (AEs) by the treating physicians | Up to 24 month study period
Identify, describe, and report any suspected AEs that occur while on treatment with Apixaban or preventing stroke and systemic embolism in patients with NVAF | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Mexico (2):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Puebla City, Puebla

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx